CLINICAL TRIAL: NCT05793021
Title: FKBP51s: a New Molecular Biomarker for Glioblastoma? Pre- and Post-operative Blood Levels Evaluation of FKBP51s Protein and Correlation With MRI Phenotype
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3751
Record Dates: First submitted 2023-02-20; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other)
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood sample pre and post surgery to determine the level of FKBP51s protein

SUMMARY:
The aim of this interventional study is to investigate the correlation between Magnetic Resonance Phenotype and levels of FKBP51s protein pre and post surgery in adult patients affected by Glioblastoma

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Diagnosis of Glioblastoma with surgery criteria
* Brain MRI with contrast both pre and post surgery

Exclusion Criteria:

* No availability of radiological documentation
* Glioblastoma diagnosis not confirmed by Histological examination
* Withdrawal of ICF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between FKBP51s protein concentration in Blood Cells and Disease flow | 1 week
Correlation between FKBP51s protein concentration in Blood Cells and Disease flow | 3 months

SECONDARY OUTCOMES:
Correlation between FKBP51s protein concentration in Blood Cells and PDL1 expression, Brain MRI phenotype and survival | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitaro "A. Gemelli" IRCCS, Roma, Italy